CLINICAL TRIAL: NCT00398398
Title: A Prospective Phase II Study of Cetuximab (Erbitux®) in Combination With XELOX [XELoda® (Capecitabine) and OXaliplatin] in Patients With Advanced Gastric Cancer
Brief Title: Study of XELOX With Cetuximab in Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0603; EMR 62202-723,OXALI_L_01600
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; chemotherapy; cetuximab; capecitabine; oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitbine, oxaliplatin, cetuximab (Experimental): Capecitbine, oxaliplatin and cetuximab every three week; Capecitabine 1,000 mg/m2 was administered twice daily on days 1-14. Oxaliplatin 130 mg/m2 i.v. for 2 h was given on day 1 after cetuximab infusion. Cetuximab at an initial loading dose of 400 mg/m2 i.v. for 2 h and, thereafter, maintenance dose of 250 mg/m2 for 1 h every week.
  Interventions: Drug: Capecitabine, Oxaliplatin, Cetuximab

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin, Cetuximab — Xelox(Capecitbine, Oxaliplatin) and Cetuximab every three week; Capecitabine 1,000 mg/m2 was administered twice daily on days 1-14. Oxaliplatin 130 mg/m2 i.v. for 2 h was given on day 1 after cetuximab infusion. Cetuximab at an initial loading dose of 400 mg/m2 i.v. for 2 h and, thereafter, maintenance dose of 250 mg/m2 for 1 h every week.
  Other Names: xeloda, oxalitin, Erbitux

SUMMARY:
The combination of capecitabine and oxaliplatin as 'backbone' regimen, adding a newer biologic agent, cetuximab, is a reasonable strategy of further chemotherapy development in advanced gastric cancer, which is the investigators study rationale.

DETAILED DESCRIPTION:
There is presently no chemotherapy regimen considered to be the global standard of care for patients with AGC, and there is still a need for new agents and/or regimens to improve the efficacy and safety of chemotherapy in advanced stomach cancers.

The combination of 5-fluorouracil plus cisplatin (FP) has been widely used for the first-line treatment of advanced gastric cancer in many countries.

Randomized phase III trial investigating capecitabine plus cisplatin(XP) versus FP showed XP is at least as good as FP with improved patients' preference.

A Phase II study of capecitabine plus oxaliplatin (XELOX) was conducted in our study group.

ELIGIBILITY:
Inclusion Criteria:

* Having given signed written informed consent
* Patients must have histologically or cytologically documented stomach adenocarcinoma including adenocarcinoma of the esophagogastric junction.
* Patients must have unresectable metastatic disease or recurrent disease after curative surgical resection with uni-dimensionally measurable disease according to RECIST (at least longest diameter 1 cm on computed tomography scan, or at least 2 cm on chest x-ray or physical examination
* Age 18 to 70 years old
* Estimated life expectancy of more than 3 months
* ECOG performance status < 2 (See Appendix E)
* Adequate bone marrow function (WBC>3,000/µL, ANC>1,500/µL, and platelets>100,000/µL, Hb>8g/dl)
* Adequate kidney function (creatinine<1.5 mg/dL)
* Adequate liver function [bilirubin< 2.0 mg/dL, transaminases levels<3 times the Upper Normal Value (5 times for patients with liver metastasis)]
* Prothrombin time not less than 50% of Lower Normal Value
* No prior chemotherapy
* No prior radiation therapy
* Patients must not have psychological, familial, sociological or geographical conditions which do not permit medical follow-up and compliance with this study.
* Women of childbearing potential must have a negative serum HCG pregnancy test on admission. Men and women of reproductive potential must have agreed to use an effective method of contraception while on treatment and for 6 months after study treatment.

Exclusion Criteria:

* Past or concurrent history of neoplasm other than gastric adenocarcinoma within the last five years, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri.
* Central nervous system (CNS) metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start
* Gastric outlet obstruction, intestinal obstruction and obvious peritoneal seeding.
* Evidence of serious gastrointestinal bleeding.
* The patient has bony lesions as the sole evaluable disease.
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception.
* Patients with sensory neuropathy (grade> 1 according to NCI CTCAE v. 3.0).
* Hypersensitivity to any of the study drugs or ingredients.
* Other serious illness or medical conditions that would not allow study participation in the best interest of the patient as decided by the investigator.
* Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry.
* History of significant neurologic or psychiatric disorders including dementia or seizures.
* Active uncontrolled infection.
* Pre-existing clinically significant diarrhea.
* Unstable diabetes mellitus.
* Severe hypercalcemia of > 12 mg/dL and uncontrolled with bisphosphonates.
* Active disseminated intravascular coagulation.
* Concurrent treatment with corticosteroids (or equivalent) except as use for the prophylactic medication regimen, treatment of acute hypersensitivity reactions or nausea, or unless chronic treatment (initiated > 6 months prior to study entry) at low dose (<20 mg methyl prednisolone or equivalent).
* Concomitant or administration of any other experimental drug under investigation within 4 weeks before the study.
* Concomitant or previous hormonal therapy, or immunotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Seoul Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Xelox Plus Cetuximab: Capecitabine, oxaliplatin and cetuximab
  cetuximab : initial loading dose of 400 mg/m2, maintenance dose of 250 mg/m2 (every week) Oxaliplatin : 130 mg/m2 (every 3 weeks) capecitabine :1,000 mg/m2 (days 1-14)
Period: Overall Study
Arm/Group | Xelox Plus Cetuximab
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Xelox Plus Cetuximab: Capecitabine, oxaliplatin and cetuximab
Arm/Group | Xelox Plus Cetuximab
Number analyzed (Participants) | 44
Age, Customized [Median (Full Range); unit: years] | 57.5 [36 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 29
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Tumor response was evaluated every two cycles by CT scans and other indicated methods, and the patients with complete or partial response required a confirmatory response evaluation at least 4 weeks later. Patients without confirmatory evaluation were not regarded as responders.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Xelox Plus Cetuximab
Number analyzed (Participants) | 44
participants | 23

2. Secondary Outcome: Progression-free Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Xelox Plus Cetuximab
Number analyzed (Participants) | 44
months | 6.5 [4.9 to 8.4]

3. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Xelox Plus Cetuximab
Number analyzed (Participants) | 44
months | 11.8 [6.7 to 16.8]

4. Secondary Outcome: Toxicity Profile
Description: Number of patients who experienced toxicity from study treatment to evaluate the safety and tolerability of XELOX plus Cetuximab
Time Frame: 1 years
Measure: Number; unit: participants
Arm/Group | Xelox Plus Cetuximab
Number analyzed (Participants) | 44
participants | 44

ADVERSE EVENTS:
Time Frame: 1 year after completion of study treatment. If patients received another treatment, toxicity assessment was not done further.
Arm/Group | Xelox Plus Cetuximab
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xelox Plus Cetuximab (N=44)
Mood disorder (Psychiatric disorders) | 1 — Mood fluctuation during treatment. But this was assessed as unlikely to be related to study treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xelox Plus Cetuximab (N=44)
Anemia (Blood and lymphatic system disorders) | 36
Leukopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Asthenia (General disorders) | 36
Anorexia (Gastrointestinal disorders) | 35
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 13
Stomatitis (Gastrointestinal disorders) | 28
Diarrhea (Gastrointestinal disorders) | 23
Sensory neuropathy (Nervous system disorders) | 33
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 34
Acneiform rash (Skin and subcutaneous tissue disorders) | 34
Abdominal pain (Gastrointestinal disorders) | 10
Elevated Aspartate aminotransferase (Hepatobiliary disorders) | 23
Elevated alanine transferase (Hepatobiliary disorders) | 16
Elevated bilirubin (Hepatobiliary disorders) | 10
Infusion reaction (Immune system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No